CLINICAL TRIAL: NCT07201623
Title: The Effect Of Web-Based Birth Preparation Education Given To Pregnant Women On Prenatal Attachment And Fear Of Birth
Acronym: Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ebru YILDIRIM, Research Assistant, Çankırı Karatekin University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E53449070-779-96
Record Dates: First submitted 2025-07-25; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Chronic Disease of Cardiovascular System
Keywords: Web-based health education; midwifery care; nursing care; birth preparation; prenatal attachment; fear of childbirth
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Materials and methods: This randomized controlled trial was conducted between February 2021 and January 2022 with the participation of 102 pregnant women who met the research criteria in family and community health centers and state hospital in Çankırı city center. Participants in the intervention group were sent 15 and 45-minute video links of the modules in the birth preparation training program uploaded to the web base. The participants' viewing status of the videos was checked weekly, and the duration of the participants in the intervention group watching the training videos for the modules was limited to 6 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): group providing web-based childbirth preparation training
  Interventions: Behavioral: web-based childbirth preparation education
- control group (No Intervention): the group that did not receive web-based childbirth preparation education

INTERVENTIONS:
Behavioral: web-based childbirth preparation education — group providing web-based childbirth preparation training
  Arms: intervention group

SUMMARY:
WEB-BASED CHILDBIRTH PREPARATION TRAINING GIVEN TO PREGNANT WOMEN PRENATAL ATTACHMENT AND ITS EFFECT ON FEAR OF CHILDBIRTH

DETAILED DESCRIPTION:
Aim: The aim of this study was to evaluate the effect of web-based childbirth preparation education on prenatal attachment and fear of childbirth.

Materials and methods: This randomized controlled trial was conducted between February 2021 and January 2022 with the participation of 102 pregnant women who met the research criteria in family and community health centers and state hospital in Çankırı city center. Participants in the intervention group were sent 15 and 45-minute video links of the modules in the birth preparation training program uploaded to the web base. The participants' viewing status of the videos was checked weekly, and the duration of the participants in the intervention group watching the training videos for the modules was limited to 6 weeks. Participants in the control group did not receive any intervention other than the routine clinical care they received. The study data were collected with a questionnaire prepared using the "Introductory Information Form", "Maternal Fetal Attachment Scale" and "Wijma Birth Expectancy Scale -A Version". The data obtained in the study were evaluated in the computer environment using the Statistical Package for the Social Sciences 22.0 statistical program.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who: · Live in Çankırı province, · 18 years of age or older, · Have no vision or hearing problems, · Have not been diagnosed with a high-risk pregnancy, · Between 28 and 32 weeks pregnant, · Able to use the internet on a computer or phone,

* Agree to be monitored via various communication tools (phone, social media), · Have not previously received childbirth preparation training or education from a pregnancy school,
* Volunteer to participate in the study were included in the study.

Exclusion Criteria:

* At each stage of the study, pregnant women who refused to participate were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Kadın cinsiyetine sahip ve gebe olanların katılımı uygundur
Enrollment: 120 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Maternal-Fetal Attachment (MFA) | 24-36 pregnancy week
  Scales have 24 five-point Likert-type items and are self-administered. The scales are scored on a scale of one to five, with five being the most positive statement. Note that the scoring is reversed for Item 22, with 'Definitely yes' scoring one point and 'Definitely no' scoring five points. The mean score is calculated by dividing the sum of the item scores by the number of items answered. Cronbach's alpha for MFA was 0.84 in Cranley's study (1981), min 2,29 max4,63 .

SECONDARY OUTCOMES:
Wijma Delivery Expectancy/Experience Questionnaire A Version (W-DEQ-A) | 28-36 pregnancy week
  The W-DEQ-A is a validated 33-item questionnaire, with scores ranging from 'not at all' (0) to 'extremely' (5), giving a minimum score of 0 and a maximum score of 165. A higher score indicates a more intense fear of childbirth.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankiri Karatekin Üniversitesi, Çankırı, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I dont know

REFERENCES:
- [Background] Ustunsoz A, Guvenc G, Akyuz A, Oflaz F. Comparison of maternal-and paternal-fetal attachment in Turkish couples. Midwifery. 2010 Apr;26(2):e1-9. doi: 10.1016/j.midw.2009.12.006. Epub 2010 Feb 20. PMID 20172635
- [Background] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- See also: Related Info — https://youtu.be/XJaBoZYvZq8